CLINICAL TRIAL: NCT03454581
Title: Comparative Effectiveness of Photobiomodulation and Manual Therapy Alone or Combined in TMD Patients: a Randomized Clinical Trial
Brief Title: Effectiveness of Photobiomodulation and Manual Therapy Alone or Combined in TMD Patients
Acronym: TMDPBMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Manoela Domingues Martins, Associate Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBM and MT TMD
Record Dates: First submitted 2018-02-05; First posted 2018-03-06 (Actual); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-08

CONDITIONS: Temporomandibular Disorder
Keywords: Temporomandibular Diseases; Photobiomodulation; Low level laser; Treatment; Manual Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Low-Level Light Therapy; phytobacteriomycin; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Photobiomodulation group (PBM) (Experimental): Gallium-aluminium-arsenide (GaAlAs) diode laser (MM Optics Recover, São Carlos, São Paulo, Brazil) with a wavelength of 808 nm, punctual contact mode,spot size of 0.03 cm2, power output of 100 mW, output density of 333 mW∕cm2, energy density of 13.3 J ∕cm2, 40 s exposure time per point, and 4 Joules (J) of total energy per point.
  18 individuals
  Interventions: Procedure: Photobiomodulation
- Manual Therapy group (MT) (Experimental): At masticatory muscles were performed circular movements, slip and compression with fingers movements. At the temporomandibular joint (TMJ) was performed a caudal distraction with anterior projection, placing the thumb on the second or third molar.
  16 individuals.
  Interventions: Procedure: Manual Therapy (MT)
- Combined therapy group (CT) (Experimental): Applied the protocols of PBM group and immediately after, to MT group. 17 individuals.
  Interventions: Procedure: Photobiomodulation; Procedure: Manual Therapy (MT)

INTERVENTIONS:
Procedure: Photobiomodulation — PBM was applied, three times a week for four consecutive weeks at 5 points in the TMJ region: superior, anterior, lateral, posterior and postero inferior to the condyle. In addition, all patients received laser application in the temporal muscle (anterior, middle and posterior), in the masseter (upper, middle and lower portion) and insertion of the medial pterygoid.
  Other Names: Low Level Laser (PBM)
  Arms: Combined therapy group (CT); Photobiomodulation group (PBM)
Procedure: Manual Therapy (MT) — Patients were submitted to MT at temporal, masseter and pterygoid medial from both sides, during 3 minutes each muscle group (Extraoral) and at masseter and lateral pterygoid (Intraoral) for 3 minutes, each total 21 minutes. MT on the TMJ region was performed for 1 minute and 3 repetitions during three times a week .
  Arms: Combined therapy group (CT); Manual Therapy group (MT)

SUMMARY:
The aim of the present study was to investigate the effect of photobiomodulation (PBM) and manual therapy (MT) isolated or combined in the reduce of pain, the improve of mandibular movements, the psychosocial aspects and the anxiety symptoms of patients with TMD.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) is a complex and multifactorial disease. Therapeutic modalities, as PBM and MT, expected to relief of symptoms, improve of function and reduce the impact of the disease in patient's life. Fifty-one TMD patients were randomly allocated to three groups: PBM group (n=18) using 808 nm, 100 milliwatt (mW), 13.3 J ∕cm2, 4 J per point), MT group (n=16) with 21 minutes sessions of MT of the masticatory muscles and TMJ and Combined Therapy group (CT) (n=17) applying the 2 protocol described above. All treatments were done three times a week for four consecutive weeks. Evaluations were performed at baseline, during the treatment (days 7, 14, 21, and 28) and follow up (day 60 and day 90). Visual analogue scale (VAS), Research Diagnostic Criteria (RDC/TMD) Axis I and II, Beck anxiety inventory (BAI) were used in different moments of evaluation time.

ELIGIBILITY:
Inclusion Criteria:

* TMD myogenic and arthrogenic diagnosis based in RDC/TMD Axis I analysis
* Pain in temporomandibular joint (TMJ)
* Limitation in mouth opening.

Exclusion Criteria:

* Current dental or physical treatment
* Polyarthritis and other rheumatic diseases
* Use of anti-inflammatory and muscle relaxant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and follow-up assessment: May 2016 to November 2016. Location: Participants were recruited from patients referred to the Department of Buco Maxillofacial Surgery and Traumatology and to the Department of Conservative Dentistry at Federal University of Rio Grande do Sul, Porto Alegre,Brazil.
Pre-assignment Details: Fifty-one participants were enrolled and randomized into 3 groups. Inclusion criteria: myogenic and arthrogenic temporomandibular dysfunction, pain and mouth movement limitation.
  Exclusion criteria: Dental therapy; rheumatic diseases, use of anti-inflammatory and muscle relaxant.
Groups:
- Photobiomodulation Group: Gallium-aluminium-arsenide (GaAlAs) diode laser (MM Optics Recover, São Carlos, São Paulo, Brazil) with a wavelength of 808 nm, punctual contact mode,spot size of 0.03 cm2, power output of 100mW (megawatts), output density of 333 mW∕cm2, energy density of 13.3 J ∕cm2, 40 s exposure time per point, and 4 Joules (J) of total energy per point.
  18 individuals
  Photobiomodulation: PBM was applied, three times a week for four consecutive weeks at 5 points in the TMJ region: superior, anterior, lateral, posterior and postero inferior to the condyle. In addition, all patients received laser application in the temporal muscle (anterior, middle and posterior), in the masseter (upper, middle and lower portion) and insertion of the medial pterygoid.
- Manual Therapy Group (MT): At masticatory muscles were performed circular movements, slip and compression with fingers movements. At the temporomandibular joint (TMJ) was performed a caudal distraction with anterior projection, placing the thumb on the second or third molar.
  16 individuals.
  Manual Therapy (MT): Patients were submitted to MT at temporal, masseter and pterygoid medial from both sides, during 3 minutes each muscle group (Extraoral) and at masseter and lateral pterygoid (Intraoral) for 3 minutes, each total 21 minutes. MT on the TMJ region was performed for 1 minute and 3 repetitions during three times a week .
- Combined Therapy Group (CT): Applied the protocols of photobiomodulation group and immediately after, to MT group.
  17 individuals.
Period: Overall Study
Arm/Group | Photobiomodulation Group | Manual Therapy Group (MT) | Combined Therapy Group (CT)
Started | 18 | 16 | 17
Completed | 14 | 13 | 14
Not Completed | 4 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Photobiomodulation Group (PBM): PBM was applied, three times a week for four consecutive weeks at 5 points in the TMJ region: superior, anterior, lateral, posterior and postero inferior to the condyle. In addition, all patients received laser application in the temporal muscle (anterior, middle and posterior), in the masseter (upper, middle and lower portion) and insertion of the medial pterygoid.
- Manual Therapy Group (MT): Patients were submitted to MT at temporal, masseter and pterygoid medial from both sides, during 3 minutes each muscle group (Extraoral) and at masseter and lateral pterygoid (Intraoral) for 3 minutes, each total 21 minutes. MT on the TMJ region was performed for 1 minute and 3 repetitions during three times a week .
- Combined Therapy Group (CT): Applied the protocols of PBM group and immediately after, to MT group.
  .
- Total: Total of all reporting groups
Arm/Group | Photobiomodulation Group (PBM) | Manual Therapy Group (MT) | Combined Therapy Group (CT) | Total
Number analyzed (Participants) | 18 | 16 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.29 (14.43) | 42.44 (17.45) | 41.65 (19.46) | 43.48 (17.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 16 | 49
  Male | 0 | 1 | 1 | 2
Duration of pain [Mean (Standard Deviation); unit: years] | 8.8 (6.9) | 10.1 (12.8) | 9.2 (9) | 9.4 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Analogic Scale (VAS) for Pain
Description: Visual Analogic Score (VAS) is a psychometric scale used to measure subjective characteristics, as pain. Consists of a 100mm horizontal line with descriptors "no pain" at the initial point (score 0) and "worst pain" at the end point (score 100). To avoid clustering of scores, numbers or verbal descriptors at intermediate points are not recommended. Patients were asked to place a handwritten mark at one point along the 100mm line that best represents their pain intensity. The scores are recorded in millimeters and determined by the measurements from the initial point of the scale to the patients' mark, using a ruler. Higher scores indicate high levels of pain intensity. In this study, the scores (mm) of pain were recorded at days 7, 14, 21, 28, 60 and 90 and compared to the baseline score (day 0) to evaluate the response to each treatment.
Time Frame: 0,7,14,21,28,60,90 days
Measure: Mean (95% Confidence Interval); unit: millimeters
Groups:
- Photobiomodulation Group: Gallium-aluminium-arsenide (GaAlAs) diode laser with a wavelength of 808 nm was applied, three times a week for four consecutive weeks at TMJ, temporal muscle, masseter and insertion of the medial pterygoid.
- Manual Therapy Group (MT): Patients were submitted to circular movements at temporal, masseter and pterygoid medial (Extraoral) and at masseter and lateral pterygoid (Intraoral) during three times a week for 4 weeks. In addition, an articular manipulation at TMJ was performed.
- Combined Therapy Group (CT): Applied the protocols of photobiomodulation group and immediately after, to MT group.
Arm/Group | Photobiomodulation Group | Manual Therapy Group (MT) | Combined Therapy Group (CT)
Number analyzed (Participants) | 14 | 13 | 14
millimeters
  Baseline | 4.1 [2.91 to 5.36] | 4.4 [2.46 to 6.31] | 5.2 [3.75 to 6.61]
  Day 7 | 3.3 [1.89 to 4.68] | 2.8 [1.51 to 4.03] | 3.4 [2.23 to 4.49]
  Day14 | 1.9 [1.10 to 2.76] | 1.7 [0.71 to 2.68] | 2.4 [1.72 to 3.13]
  Day 21 | 1.8 [0.77 to 2.8] | 0.5 [0.03 to 1.04] | 1.9 [1.12 to 2.59]
  Day 28 | 1.1 [0.43 to 1.71] | 1.3 [0.17 to 2.44] | 0.9 [0.43 to 1.43]
  Day 60 | 0.8 [0.19 to 1.39] | 0.6 [0.16 to 1.07] | 1.2 [0.72 to 1.71]
  Day 90 | 1.6 [0.96 to 2.27] | 0.9 [0.17 to 1.66] | 1.9 [0.79 to 2.92]
Statistical Analysis 1: Comparison: Photobiomodulation Group vs Manual Therapy Group (MT) vs Combined Therapy Group (CT); Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Final Values) = 0.05

2. Secondary Outcome: Change at Jaw Movements
Description: Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) Axis I was used to provide information of jaw movements. Using a caliper to assess mandibular range of motion (in millimeters), we measure mouth opening, right and left deviations and protrusion.
  This questionnaire was applied at baseline (day 0), end of the treatment (day 28) and follow up (day 90).
Time Frame: 0,28,90 days
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Photobiomodulation Group | Manual Therapy Group (MT) | Combined Therapy Group (CT)
Number analyzed (Participants) | 14 | 13 | 14
millimeters
  Opening - Day 0 | 29.64 [27.17 to 32.35] | 27.92 [24.97 to 31.23] | 29.71 [25.49 to 34.64]
  Opening - Day 28 | 35.27 [29.53 to 35.92] | 34.00 [30.85 to 37.47] | 31.50 [29.27 to 33.90]
  Opening - Day 90 | 36.86 [34.51 to 39.36] | 33.38 [30.78 to 36.21] | 31.93 [30.41 to 33.52]
  Maximum opening - day 0 | 40.86 [37.62 to 44.09] | 38.46 [35.06 to 41.86] | 35.29 [31.02 to 39.54]
  Maximum opening - day 28 | 42.79 [40.15 to 45.42] | 41.85 [39.60 to 44.09] | 38.93 [36.70 to 41.16]
  Maximum opening - day 90 | 44.50 [42.24 to 46.76] | 42.54 [39.56 to 45.51] | 39.93 [37.86 to 42.00]
  Right excursion - day 0 | 5.93 [4.26 to 8.26] | 6.31 [5.13 to 7.76] | 6.57 [5.21 to 8.29]
  Right excursion - day 28 | 8.36 [7.21 to 9.68] | 8.62 [6.91 to 10.74] | 6.64 [5.63 to 7.83]
  Right excursion - day 90 | 7.90 [6.69 to 9.33] | 8.31 [7.06 to 9.78] | 7.36 [6.57 to 8.24]
Statistical Analysis 1: Comparison: Photobiomodulation Group vs Manual Therapy Group (MT) vs Combined Therapy Group (CT); Test type: Superiority or Other; p = 0.05, Generalized Estimating Equation

3. Secondary Outcome: Change on Chronic Pain Grades
Description: RDC/TMD Axis II includes measures from the Graded Chronic Pain Scale (GCPS). Participants rated on scales from 0 = "no pain" to 10 = "pain as bad as could be" their current pain and average and worst facial pain in the past six months. Also, on scales from 0 = "no interference" to 10 = "unable to carry on any activities" the degree of facial pain interference with daily activities in the past six months. The mean of the ratings, multiplied by 10, gives information on characteristic pain intensity (CPI) and daily disability. The GCP is based on CPI, number of disability days in the past six months and daily disability score classified as 0 = no pain, I = low CPI and disability, II = high CPI and low pain-related disability, III = moderate CPI and disability, and IV = severe CPI and disability. In this study, the number of participants, at the end of the study, with Low Incapacity (Grades 0 to I) and Higher Incapacity (Grades II to IV) was compared to the baseline numbers.
Time Frame: 0,90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Photobiomodulation Group | Manual Therapy Group (MT) | Combined Therapy Group (CT)
Number analyzed (Participants) | 14 | 13 | 14
Participants
  Day 0: Low Incapacity | 10 | 12 | 7
  Day 0: High Incapacity | 4 | 1 | 7
  Day 90: Low Incapacity | 13 | 13 | 8
  Day 90: High Incapacity | 1 | 0 | 6
Statistical Analysis 1: Comparison: Photobiomodulation Group vs Manual Therapy Group (MT) vs Combined Therapy Group (CT); Test type: Superiority or Other; p = 0.05, Generalized Estimating Equation

4. Secondary Outcome: Changes on Levels of Depression Symptoms
Description: RDC/TMD Axis II is a validated questionnaire which assess the levels of depression symptoms (LDS). The participants answered 20 questions about how much they have been distressed to several symptoms of depression rating on a scale: 0 =Not at all; 1= A little bit; 2=Moderately; 3=Quite a bit; 4=Extremely. The total number of participants in the end of study, with no depression (scores 0 and 1 on the scale) and with moderate and severe depression (scores 2 to 4 on the scale) was compared to the baseline numbers (day 0).
Time Frame: 0,90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Photobiomodulation Group | Manual Therapy Group (MT) | Combined Therapy Group (CT)
Number analyzed (Participants) | 14 | 13 | 14
Participants
  Day 0: No depression | 6 | 7 | 3
  Day 0: Moderate/Severe depression | 8 | 6 | 11
  Day 90: No depression | 11 | 9 | 9
  Day 90: Moderate/Severe depression | 3 | 4 | 5
Statistical Analysis 1: Comparison: Photobiomodulation Group vs Manual Therapy Group (MT) vs Combined Therapy Group (CT); Test type: Superiority or Other; p < 0.05, Generalized Estimating Equation

5. Secondary Outcome: Change on Nonspecific Physical Symptoms With Pain
Description: RDC/TMD Axis II can be used to provide information on nonspecific physical symptoms with pain. The participants rate the experiences in the past few weeks relative to "how usually feels" about several pain symptoms as follows: 0 =Not at all; 1= A little bit; 2=Moderately; 3=Quite a bit; 4=Extremely. We divided the participants into no symptoms ("Normal" = scores 0 to1 at the scale) and moderate/severe symptoms (scale 2 to 4 at the scale) and compared the total number of participants in each classification (No symptoms and Moderate/severe symptoms) at the end of the study to the baseline numbers.
Time Frame: 0, 90 days
Measure: Count of Participants; unit: Participants
Groups:
- Combined Therapy Group (CT): Applied the protocols of photobiomodulation group and immediately after, to MT group.
  .
Arm/Group | Photobiomodulation Group | Manual Therapy Group (MT) | Combined Therapy Group (CT)
Number analyzed (Participants) | 14 | 13 | 14
Participants
  Day 0: Normal | 3 | 5 | 2
  Day 0: Moderate/Severe symptoms | 11 | 8 | 12
  Day 90: Normal | 7 | 10 | 6
  Day 90: Moderate/Severe symptoms | 7 | 3 | 8
Statistical Analysis 1: Comparison: Photobiomodulation Group vs Manual Therapy Group (MT) vs Combined Therapy Group (CT); Test type: Other; p < 0.01, Generalized Estimating Equation

6. Secondary Outcome: Change on Nonspecific Physical Symptoms Without Pain
Description: RDC/TMD Axis II is also used to provide information on nonspecific physical symptoms without pain. The participants rate the experiences in the past few weeks relative to "how usually feels" about several symptoms nonrelated to pain as follows: 0 =Not at all; 1= A little bit; 2=Moderately; 3=Quite a bit; 4=Extremely. We divided the participants in no symptoms ("Normal" =scores 0 to1 at the scale) and moderate/severe symptoms (scale 2 to 4 at the scale) and compared the total number of participants in each classification at the end of the study to the baseline numbers.
Time Frame: 0, 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Photobiomodulation Group | Manual Therapy Group (MT) | Combined Therapy Group (CT)
Number analyzed (Participants) | 14 | 13 | 14
Participants
  Day 0: Normal | 5 | 6 | 2
  Day 0: Moderate/Severe symptoms | 9 | 7 | 12
  Day 90: Normal | 8 | 11 | 8
  Day 90: Moderate/Severe symptoms | 6 | 2 | 6
Statistical Analysis 1: Comparison: Photobiomodulation Group vs Manual Therapy Group (MT) vs Combined Therapy Group (CT); Test type: Superiority or Other; p = 0.05, Generalized Estimating Equation

7. Secondary Outcome: Changes on Mandibular Function
Description: The changes at mandibular functions can be evaluated using the question 19 of RDC/TMD Axis II. Participants answered 0=No (no limitation due to jaw problem) or 1=Yes (the activity is limited by the jaw problem - worse outcome) to a list of activities that the jaw problem can limit from doing. The mean of all the "Yes" answers (score 1) for each group in the end of the study (day 90) was calculated and compared to the baseline means.
Time Frame: 0, 90 days
Population: To the Analysis of Population, we used the mean and the confidence interval of scores of all participants from each group.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Photobiomodulation Group | Manual Therapy Group (MT) | Combined Therapy Group (CT)
Number analyzed (Participants) | 14 | 13 | 14
score on a scale
  Chewing - day 0 | 0.5 [0.26 to 0.74] | 0.85 [0.55 to 0.96] | 0.93 [0.63 to 0.99]
  Chewing - day 90 | 0.29 [0.11 to 0.56] | 0.38 [0.17 to 0.66] | 0.57 [0.32 to 0.79]
  Exercising - day 0 | 0.07 [0.01 to 0.37] | 0.08 [0.01 to 0.39] | 0.50 [0.26 to 0.74]
  Exercising - day 90 | 0.00 [0.00 to 0.00] | 0.08 [0.01 to 0.39] | 0.07 [0.01 to 0.37]
  Eating hard foods - day 0 | 0.71 [0.44 to 0.89] | 0.85 [0.55 to 0.96] | 0.36 [0.16 to 0.62]
  Eating hard foods - day 90 | 0.43 [0.21 to 0.68] | 0.54 [0.28 to 0.78] | 0.71 [0.44 to 0.89]
  Eating soft foods - day 0 | 0.07 [0.01 to 0.37] | 0.23 [0.08 to 0.52] | 0.36 [0.16 to 0.62]
  Eating soft foods - day 90 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.14 [0.04 to 0.43]
  Smiling - day 0 | 0.36 [0.16 to 0.62] | 0.31 [0.12 to 0.59] | 0.50 [0.26 to 0.74]
  Smiling - day 90 | 0.07 [0.01 to 0.37] | 0.08 [0.01 to 0.39] | 0.36 [0.16 to 0.62]
  Swallowing - day 0 | 0.14 [0.04 to 0.43] | 0.23 [0.08 to 0.52] | 0.43 [0.21 to 0.68]
  Swallowing - day 90 | 0.07 [0.01 to 0.37] | 0.00 [0.00 to 0.00] | 0.21 [0.07 to 0.49]
Statistical Analysis 1: Comparison: Photobiomodulation Group vs Manual Therapy Group (MT) vs Combined Therapy Group (CT); Test type: Superiority or Other; p = 0.05, Generalized Estimating Equation

8. Secondary Outcome: Changes on Levels of Anxiety
Description: Beck anxiety inventory (BAI) is a validated questionnaire with 21 multiple-choice items addressing how much the patient has been bothered by common symptoms of anxiety, at the list in the previous week. Each answer is scored on a scale value of 0 = not at all , 1=Mildly, but it didn't bother me much, 2=Moderately - it wasn't pleasant at times and 3=Severely - it bothered me a lot. We applied the BAI in two moments of the study (baseline and at follow -up= day 90). In each moment the participants were classified using a score calculated by finding the sum of the 21 items. Score of 0-21 = low anxiety, Score of 22-35 = moderate anxiety, Score of 36 and above = high levels of anxiety. We presented the results using only the mean of BAI of participants of each group in that moment. We compared the mean of BAI among the groups (PBM X MT X combined groups- intergroup analysis) in the baseline and follow-up period. In addition, we also analyzed intragroup results comparing the mean of BAI.
Time Frame: 0,90 days
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Photobiomodulation Group | Manual Therapy Group (MT) | Combined Therapy Group (CT)
Number analyzed (Participants) | 14 | 13 | 14
score on a scale
  Day 0 | 17.86 [8.56 to 27.15] | 14.92 [6.31 to 23.54] | 31.21 [21.93 to 40.49]
  Day 90 | 9.57 [2.01 to 17.14] | 7.92 [3.93 to 11.91] | 13.57 [8.54 to 18.60]
Statistical Analysis 1: Comparison: Photobiomodulation Group vs Manual Therapy Group (MT) vs Combined Therapy Group (CT); Test type: Superiority or Other; p = 0.05, Generalized Estimating Equation

ADVERSE EVENTS:
Groups:
- Photobiomodulation Group (PBM): Gallium-aluminium-arsenide (GaAlAs) diode laser with a wavelength of 808 nm was applied, three times a week for four consecutive weeks at TMJ, temporal muscle, masseter and insertion of the medial pterygoid.
- Combined Therapy Group (CT): Applied the protocols of PBM group and immediately after, to MT group.
Arm/Group | Photobiomodulation Group (PBM) | Manual Therapy Group (MT) | Combined Therapy Group (CT)
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No